CLINICAL TRIAL: NCT06268873
Title: A Phase III, Randomised, Double-Blind Study to Assess the Efficacy, Safety and Tolerability of Baxdrostat in Combination With Dapagliflozin Compared With Dapagliflozin Alone on Chronic Kidney Disease (CKD) Progression in Participants With CKD and High Blood Pressure
Brief Title: A Phase III Study to Investigate the Efficacy and Safety of Baxdrostat in Combination With Dapagliflozin on CKD Progression in Participants With CKD and High Blood Pressure.
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D6972C00003; 2023-506457-38-00 (Registry Identifier: EU CT number)
Record Dates: First submitted 2024-02-13; First posted 2024-02-20 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Chronic Kidney Disease and Hypertension
Keywords: Chronic kidney disease; Hypertension; Blood pressure; Baxdrostat; Dapagliflozin
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Baxdrostat/dapagliflozin (Experimental): Participants randomised to the baxdrostat/dapagliflozin arm will initially receive a dose of baxdrostat lower dose and dapagliflozin. For participants that meet the up-titration criteria, baxdrostat may be up-titrated to higher dose.
  Interventions: Drug: Baxdrostat/dapagliflozin
- Dapagliflozin (Active Comparator): Patients will receive one dose of dapagliflozin (active comparator) in combination with placebo matching baxdrostat daily
  Interventions: Drug: Dapagliflozin in combination with placebo

INTERVENTIONS:
Drug: Baxdrostat/dapagliflozin — baxdrostat tablet
  dapagliflozin tablet
  Other Names: Baxdrostat CIN-107
  Arms: Baxdrostat/dapagliflozin
Drug: Dapagliflozin in combination with placebo — dapagliflozin tablet
  placebo tablet
  Arms: Dapagliflozin

SUMMARY:
The purpose of this study is to measure the efficacy and safety of baxdrostat/dapagliflozin in participants ≥ 18 years of age with CKD and HTN.

This study consists of a screening, a 4-week dapagliflozin run-in period for participants untreated with SGLT2i at baseline; a 24-month double-blind period in which participants will receive either baxdrostat/dapagliflozin or placebo/dapagliflozin; and approximately 12-week open-label period in which all participants will discontinue baxdrostat/placebo and receive dapagliflozin alone. Site visits will take place at 2-, 4-, 8-, and 16- weeks following randomisation. Thereafter visits will occur approximately every 4 months, until the 24-month visit at which time baxdrostat/placebo will be discontinued. Participants will continue open-label dapagliflozin for another 12-weeks (approximately), where reassessment of eGFR will occur for the primary efficacy endpoint.

In the event of premature discontinuation of blinded study intervention, participants will continue in the study and receive open-label dapagliflozin monotherapy, unless the participant meets dapagliflozin specific discontinuation criteria, in which case all study interventions will be discontinued.

ELIGIBILITY:
Inclusion Criteria:

1. Participants of any sex and gender must be ≥ 18 years old, or older, at the time of signing the informed consent.
2. Participants with CKD and eGFR ≥ 30 and < 90 mL/min/1.73 m2 at screening
3. Urine albumin creatinine ratio > 200 mg/g (22.6 mg/mmol) and < 5000 mg/g (565 mg/mmol) at screening
4. Participants with history of HTN and a SBP ≥ 130 mmHg at screening and ≥ 120 mmHg at the randomisation visit
5. Stable and maximum tolerated dose of an ACE inhibitor or an ARB (not both) for at least 4 weeks prior to Screening Visit
6. Central laboratory serum potassium must meet the following criteria at the Screening Visit, based on screening eGFR:

   * for participants with screening eGFR ≥ 45 mL/min/1.73 m2, potassium must be ≥ 3.0 and ≤ 4.8 mmol/L at the Screening Visit
   * for participants with screening eGFR < 45 mL/min/1.73 m2, potassium must be ≥ 3.0 and ≤ 4.5 mmol/L at the Screening Visit

Exclusion Criteria:

1. Systolic blood pressure > 180 mmHg, or DBP > 110 mmHg at screening.
2. Known hyperkalaemia, defined as potassium of ≥ 5.5 mmol/L within 3 months at screening.
3. Serum sodium < 135 mmol/L at the Screening Visit, determined as per central laboratory.
4. Diabetes mellitus:

   (a) T1DM at Screening Visit: (i) For US only: patients with T1DM treated with SGLT2i for at least 4 months, without DKA during that period, and who have experience with ketone monitoring are eligible for inclusion.

   (ii) For Japan only: patients with T1DM treated with dapagliflozin 10 mg for at least 4 months, without DKA during the period of dapagliflozin treatment are eligible for inclusion.

   (b) Uncontrolled T2DM at screening: HbA1C > 10.5% (> 91 mmol/mol).
5. New York Heart Association functional HF class IV at screening.
6. Stroke, transient ischaemic cerebral attack, valve implantation or valve replacement, carotid surgery, or carotid angioplasty, acute coronary syndrome, or hospitalisation for worsening heart failure within previous 3 months prior to randomisation.
7. Any dialysis (including for acute kidney injury) within 3 months prior to Screening Visit.
8. Any acute kidney injury within 3 months prior to the Screening Visit
9. History of organ transplant or bone marrow transplant, or planned organ transplant within 6 months following randomisation (including kidney transplant).
10. History or ongoing allergy/hypersensitivity, as judged by the investigator, to SGLT2 inhibitor (eg, empagliflozin) or ASI.
11. Any clinical condition requiring systemic immunosuppression therapy other than stable maintenance therapy for at least 3 months prior to Visit 1.
12. Any use of mineralocorticoid receptor antagonists (such as spironolactone, eplerenone, or finerenone), potassium-sparing diuretics (such as triamterene or amiloride), or potassium binders (such as sodium zirconium cyclosilicate, patiromer, or sodium polystyrene sulfonate) within 4 weeks prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2554 (Actual)
Dates: Start 2024-03-29 (Actual); Primary Completion 2028-02-24 (Estimated); Study Completion 2028-02-24 (Estimated)

PRIMARY OUTCOMES:
To determine whether baxdrostat/dapagliflozin is superior to dapagliflozin alone to slow CKD progression, assessed as the effect on change in eGFR over time. | Baseline - 2 years + 12 weeks
  Change from baseline in eGFR to post treatment.

SECONDARY OUTCOMES:
To determine whether baxdrostat/dapagliflozin is superior to dapagliflozin alone at reducing UACR (urine albumin-creatinine ratio). | Baseline -16 weeks
  Change from baseline in UACR
To determine whether baxdrostat/dapagliflozin is superior to dapagliflozin alone at reducing SBP. | Baseline -16 weeks
  Change from baseline in systolic BP (blood pressure).
To determine whether baxdrostat/dapagliflozin compared with dapagliflozin alone slows CKD progression and reduces the risk of ESKD (End-stage kidney disease). | baseline - 2 years + 12 weeks
  Kidney hierarchical composite endpoint.*
  *Defined as the most severe outcome of the following: 1. Death; 2. KFRT (chronic dialysis or kidney transplant); 3. Sustained GFR < 15 mL/min/1.73 m2; 4. Sustained GFR decline from baseline of ≥ 57%; 5 Sustained GFR decline from baseline of ≥ 50%; or 6. individual change from baseline to post-treatment eGFR if none of the outcomes occurred.
To determine whether baxdrostat/dapagliflozin compared with dapagliflozin alone slows the rate of kidney function decline after the hemodynamically-mediated acute effect on GFR (Glomerular Filtration Rate). | 8 weeks following randomisation to end of treatment
  Change in eGFR from following randomisation.
To determine whether baxdrostat/dapagliflozin is superior to dapagliflozin alone in reducing the risk of MACE | Baseline - 24 months
  Time to the first occurrence of any of the components of the composite of:
  1. CV death
  2. HF with and without hospitalization
  3. MI
  4. Stroke

OTHER OUTCOMES:
Adverse Events - Number of participants with Adverse Events | Baseline - 24 months
Clinical Laboratory - Number of participants with Abnormal clinical laboratory measurements | Baseline - 24 months
Vital Signs - Number of participants with Abnormal vital signs | Baseline - 24 months
Electrocardiogram- Number of Participants With Abnormal ECG | Baseline - 24 months

CONTACTS AND LOCATIONS:
Locations (473):
- United States (98):
  - Research Site, Fairhope, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Surprise, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Searcy, Arkansas
  - Research Site, Beverly Hills, California
  - Research Site, Canyon Country, California
  - Research Site, Fremont, California
  - Research Site, Fullerton, California
  - Research Site, Lincoln, California
  - Research Site, Los Alamitos, California
  - Research Site, San Francisco, California
  - Research Site, Stanford, California
  - Research Site, Tarzana, California
  - Research Site, Arvada, Colorado
  - Research Site, Denver, Colorado
  - Research Site, New Britain, Connecticut
  - Research Site, Boca Raton, Florida
  - Research Site, Boynton Beach, Florida
  - Research Site, Edgewater, Florida
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Hollywood, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Lake City, Florida
  - Research Site, Lake Worth, Florida
  - Research Site, Melbourne, Florida
  - Research Site, Miami, Florida
  - Research Site, Miami Lakes, Florida
  - Research Site, New Port Richey, Florida
  - Research Site, Ocoee, Florida
  - Research Site, Orlando, Florida
  - Research Site, Port Charlotte, Florida
  - Research Site, Port Orange, Florida
  - Research Site, Riverview, Florida
  - Research Site, Winter Haven, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Conyers, Georgia
  - Research Site, Macon, Georgia
  - Research Site, Champaign, Illinois
  - Research Site, Hazel Crest, Illinois
  - Research Site, Huntley, Illinois
  - Research Site, Rockford, Illinois
  - Research Site, Evansville, Indiana
  - Research Site, Fort Wayne, Indiana
  - Research Site, Hutchinson, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, Bethesda, Maryland
  - Research Site, Lanham, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, New Bedford, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Pontiac, Michigan
  - Research Site, Saint Joseph, Michigan
  - Research Site, City of Saint Peters, Missouri
  - Research Site, Kansas City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Eatontown, New Jersey
  - Research Site, Binghamton, New York
  - Research Site, Manhasset, New York
  - Research Site, Middletown, New York
  - Research Site, New York, New York
  - Research Site, Niagara Falls, New York
  - Research Site, Orchard Park, New York
  - Research Site, Rockville Centre, New York
  - Research Site, Greenville, North Carolina
  - Research Site, Jacksonville, North Carolina
  - Research Site, New Bern, North Carolina
  - Research Site, Statesville, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Columbus, Ohio
  - Research Site, Maumee, Ohio
  - Research Site, Chester, Pennsylvania
  - Research Site, Langhorne, Pennsylvania
  - Research Site, Uniontown, Pennsylvania
  - Research Site, East Providence, Rhode Island
  - Research Site, Providence, Rhode Island
  - Research Site, Charleston, South Carolina
  - Research Site, Columbia, South Carolina
  - Research Site, Sioux Falls, South Dakota
  - Research Site, Chattanooga, Tennessee
  - Research Site, Memphis, Tennessee
  - Research Site, Arlington, Texas
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Humble, Texas
  - Research Site, Lewisville, Texas
  - Research Site, Odessa, Texas
  - Research Site, Pasadena, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Burlington, Vermont
  - Research Site, Arlington, Virginia
  - Research Site, Manassas, Virginia
  - Research Site, Newport News, Virginia
  - Research Site, Salem, Virginia
  - Research Site, Woodbridge, Virginia
- Argentina (10):
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, Ciudad Autonoma de Bs As
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Córdoba
  - Research Site, La Plata
  - Research Site, Lanús
  - Research Site, Mar del Plata
  - Research Site, Mendoza
  - Research Site, San Nicolás
- Australia (8):
  - Research Site, Birtinya
  - Research Site, Clayton
  - Research Site, Darlinghurst
  - Research Site, Gosford
  - Research Site, Kogarah
  - Research Site, Perth
  - Research Site, St Leonards
  - Research Site, Wollongong
- Belgium (10):
  - Research Site, Aalst
  - Research Site, Bonheiden
  - Research Site, Brussels
  - Research Site, Ghent
  - Research Site, Ieper
  - Research Site, Kortrijk
  - Research Site, Leuven
  - Research Site, Liège
  - Research Site, Roeselare
  - Research Site, Ronse
- Brazil (10):
  - Research Site, Belém
  - Research Site, Campina Grande do Sul
  - Research Site, Campinas
  - Research Site, Curitiba
  - Research Site, Fortaleza
  - Research Site, Joinville
  - Research Site, Maringá
  - Research Site, Porto Alegre
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
- Bulgaria (11):
  - Research Site, Dupnitsa
  - Research Site, Gotse Delchev
  - Research Site, Kozloduy
  - Research Site, Lom
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Sandanski
  - Research Site, Sliven
  - Research Site, Stara Zagora
  - Research Site, Veliko Tarnovo
  - Research Site, Yambol
- Canada (17):
  - Research Site, Edmonton, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, Halifax, Nova Scotia
  - Research Site, Sydney, Nova Scotia
  - Research Site, Brampton, Ontario
  - Research Site, Concord, Ontario
  - Research Site, London, Ontario
  - Research Site, Oshawa, Ontario
  - Research Site, Stoney Creek, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Waterloo, Ontario
  - Research Site, Laval, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Sherbrooke, Quebec
  - Research Site, Saint John
- Chile (4):
  - Research Site, Araucania
  - Research Site, Santiago
  - Research Site, Valdivia
  - Research Site, Victoria
- China (33):
  - Research Site, Baotou
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Changzhou
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Dongguan
  - Research Site, Foshan
  - Research Site, Guangzhou
  - Research Site, Guiyang
  - Research Site, Haikou
  - Research Site, Hangzhou
  - Research Site, Hengyang
  - Research Site, Huai'an
  - Research Site, Lanzhou
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Ningbo
  - Research Site, Panjin
  - Research Site, Pingxiang
  - Research Site, Sanya
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Shenzhen
  - Research Site, Ürümqi
  - Research Site, Wuhan
  - Research Site, Wuxi
  - Research Site, Xi'an
  - Research Site, Xiamen
  - Research Site, Yantai
  - Research Site, Yinchuan
  - Research Site, Zhengzhou
- Czechia (8):
  - Research Site, Frýdek-Místek
  - Research Site, Jilemnice
  - Research Site, Krnov
  - Research Site, Náchod
  - Research Site, Olomouc
  - Research Site, Police nad Metují
  - Research Site, Prague
  - Research Site, Třebíč
- Denmark (7):
  - Research Site, Aalborg
  - Research Site, Aarhus
  - Research Site, Copenhagen E
  - Research Site, Esbjerg
  - Research Site, Herlev
  - Research Site, Herning
  - Research Site, Holbæk
- France (20):
  - Research Site, Amiens
  - Research Site, Annonay
  - Research Site, Bois-Guillaume
  - Research Site, Bordeaux
  - Research Site, Boulogne-Billancourt
  - Research Site, Brest
  - Research Site, Clermont-Ferrand
  - Research Site, La Roche-sur-Yon
  - Research Site, Le Puy-en-Velay
  - Research Site, Lille
  - Research Site, Marseille
  - Research Site, Nîmes
  - Research Site, Paris
  - Research Site, Poitiers
  - Research Site, Quimper
  - Research Site, Sarcelles
  - Research Site, Toulouse
  - Research Site, Tours
  - Research Site, Valenciennes
  - Research Site, Vandœuvre-lès-Nancy
- Germany (19):
  - Research Site, Aachen
  - Research Site, Amberg
  - Research Site, Bad Oeynhausen
  - Research Site, Berlin
  - Research Site, Bochum
  - Research Site, Dresden
  - Research Site, Essen
  - Research Site, Falkensee
  - Research Site, Hamburg
  - Research Site, Herne
  - Research Site, Leipzig
  - Research Site, Mainz
  - Research Site, München
  - Research Site, Münster
  - Research Site, Nuremberg
  - Research Site, Oldenburg
  - Research Site, Reinfeld (Holstein)
  - Research Site, Ulm
  - Research Site, Völklingen
- Greece (6):
  - Research Site, Alexandroupoli
  - Research Site, Athens
  - Research Site, Heraklion
  - Research Site, Ioannina
  - Research Site, Pátrai
  - Research Site, Thessaloniki
- Hungary (7):
  - Research Site, Békéscsaba
  - Research Site, Budapest
  - Research Site, Kecskemét
  - Research Site, Nyíregyháza
  - Research Site, Pécs
  - Research Site, Siófok
  - Research Site, Székesfehérvár
- India (12):
  - Research Site, Bangalore
  - Research Site, Belagavi
  - Research Site, Calicut
  - Research Site, Chennai
  - Research Site, Coimbatore
  - Research Site, Dehradun
  - Research Site, Hyderabad
  - Research Site, Kolkata
  - Research Site, Madurai
  - Research Site, New Delhi
  - Research Site, Pune
  - Research Site, Vijayawada
- Israel (8):
  - Research Site, Ashkelon
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Petah Tikva
  - Research Site, Ramat Gan
  - Research Site, Rehovot
  - Research Site, Tel Aviv
- Italy (10):
  - Research Site, Bologna
  - Research Site, Catanzaro
  - Research Site, Chiavari
  - Research Site, Desio
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Parma
  - Research Site, Rozzano
  - Research Site, San Giovanni Rotondo
  - Research Site, Torino
- Japan (34):
  - Research Site, Chūōku
  - Research Site, Daito-shi
  - Research Site, Fujisawa-shi
  - Research Site, Fukuoka
  - Research Site, Hiroshima
  - Research Site, Ina-shi
  - Research Site, Kamakura-shi
  - Research Site, Kasugai-shi
  - Research Site, Kawaguchi
  - Research Site, Kofu
  - Research Site, Kumagaya-shi
  - Research Site, Kurume-shi
  - Research Site, Kyoto
  - Research Site, Marugame-shi
  - Research Site, Matsuyama
  - Research Site, Nagoya
  - Research Site, Naka
  - Research Site, Nishinomiya-Shi
  - Research Site, Obihiro-shi
  - Research Site, Osaka
  - Research Site, Ōita
  - Research Site, Sakaishi
  - Research Site, Sapporo
  - Research Site, Sendai
  - Research Site, Shinjyuku-ku
  - Research Site, Shizuoka
  - Research Site, Takatsuki-shi
  - Research Site, Toride-shi
  - Research Site, Toyota-Shi
  - Research Site, Tsu
  - Research Site, Ueda-shi
  - Research Site, Urayasu
  - Research Site, Yaizu-shi
  - Research Site, Yokohama
- Malaysia (6):
  - Research Site, Klang
  - Research Site, Kota Kinabalu
  - Research Site, Kuala Lumpur
  - Research Site, Kuantan
  - Research Site, Seremban
  - Research Site, Taiping
- Netherlands (7):
  - Research Site, Alkmaar
  - Research Site, Amersfoort
  - Research Site, Dordrecht
  - Research Site, Hardenberg
  - Research Site, Harderwijk
  - Research Site, Hilversum
  - Research Site, Utrecht
- Peru (4):
  - Research Site, Arequipa
  - Research Site, Chorrillos
  - Research Site, Lima
  - Research Site, Piura
- Philippines (6):
  - Research Site, Cebu City
  - Research Site, Davao City
  - Research Site, Iloilo City
  - Research Site, Laguna
  - Research Site, Manila
  - Research Site, Quezon City
- Poland (13):
  - Research Site, Chrzanów
  - Research Site, Gdynia
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Olsztyn
  - Research Site, Poznan
  - Research Site, Rzeszów
  - Research Site, Szczecin
  - Research Site, Tczew
  - Research Site, Warsaw
  - Research Site, Wroclaw
  - Research Site, Żywiec
- Romania (6):
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Iași
  - Research Site, Oradea
  - Research Site, Târgu Mureş
  - Research Site, Timișoara
- Saudi Arabia (2):
  - Research Site, Dammam
  - Research Site, Riyadh
- Serbia (4):
  - Research Site, Belgrade
  - Research Site, Kragujevac
  - Research Site, Niš
  - Research Site, Novi Sad
- Slovakia (10):
  - Research Site, Banská Bystrica
  - Research Site, Lučenec
  - Research Site, Martin
  - Research Site, Myjava
  - Research Site, Nitra
  - Research Site, Prešov
  - Research Site, Púchov
  - Research Site, Rožňava
  - Research Site, Trnava
  - Research Site, Žilina
- South Africa (8):
  - Research Site, Benoni
  - Research Site, Cape Town
  - Research Site, Durban
  - Research Site, KwaDukuza
  - Research Site, Lenasia
  - Research Site, Midrand
  - Research Site, Newton
  - Research Site, Parow
- South Korea (11):
  - Research Site, Ansan-si
  - Research Site, Anyang-si
  - Research Site, Busan
  - Research Site, Cheonan-si
  - Research Site, Daejeon
  - Research Site, Goyang-si
  - Research Site, Gwangju
  - Research Site, Seoul
  - Research Site, Uijeongbu-si
  - Research Site, Wŏnju
  - Research Site, Yangsan
- Spain (11):
  - Research Site, A Coruña
  - Research Site, Almería
  - Research Site, Badalona
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Lugo
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Palma deMallorca
  - Research Site, Pamplona
  - Research Site, Seville
  - Research Site, Valencia
- Sweden (7):
  - Research Site, Danderyd
  - Research Site, Gävle
  - Research Site, Gothenburg
  - Research Site, Linköping
  - Research Site, Rättvik
  - Research Site, Stockholm
  - Research Site, Uppsala
- Taiwan (6):
  - Research Site, Kaohsiung City
  - Research Site, New Taipei City
  - Research Site, Taichung
  - Research Site, Taipei
  - Research Site, Taoyuan District
  - Research Site, Yung Kang City
- Thailand (7):
  - Research Site, Bangkok
  - Research Site, Chiang Mai
  - Research Site, Hat Yai
  - Research Site, Muang
  - Research Site, Phutthamonthon
  - Research Site, Ratchathewi
  - Research Site, Ubonratchathani
- Turkey (Türkiye) (10):
  - Research Site, Adana
  - Research Site, Adapazarı
  - Research Site, Afyonkarahisar
  - Research Site, Ankara
  - Research Site, Antalya
  - Research Site, Bursa
  - Research Site, Istanbul
  - Research Site, Kahramanmaraş
  - Research Site, Kayseri
  - Research Site, Kocaeli
- Ukraine (6):
  - Research Site, Chernivtsі
  - Research Site, Ivano-Frankivsk
  - Research Site, Kyiv
  - Research Site, Ternopil
  - Research Site, Uzhhorod
  - Research Site, Vinnytsia
- United Kingdom (12):
  - Research Site, Bristol
  - Research Site, Cambridge
  - Research Site, Dundee
  - Research Site, Glasgow
  - Research Site, Harrow
  - Research Site, Hounslow
  - Research Site, Leicester
  - Research Site, Liverpool
  - Research Site, London
  - Research Site, Newcastle-under-Lyme
  - Research Site, Nottingham
  - Research Site, Wolverhampton
- Vietnam (5):
  - Research Site, Can Tho
  - Research Site, Da Nang
  - Research Site, Haiphong
  - Research Site, Ho Chi Minh City
  - Research Site, Hochiminh City

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- [Derived] Dwyer JP, Maklad N, Vedin O, Monyak J, Myte R, Chertow GM, Heerspink HJL, Little DJ. Efficacy and Safety of Baxdrostat in Participants with CKD and Uncontrolled Hypertension: A Randomized, Double-Blind, Placebo-Controlled Trial. J Am Soc Nephrol. 2025 Sep 6. doi: 10.1681/ASN.0000000849. Online ahead of print. No abstract available. PMID 40913594